CLINICAL TRIAL: NCT05727501
Title: Comparison of Post Isometric Relaxation and Post Facilitation Stretching on Hamstring Muscle Flexibility in Collegiate Athletes
Brief Title: Comparison of Post Isometric Relaxation and Post Facilitation Stretching on Hamstring Muscle Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zohaibahmad0442
Record Dates: First submitted 2023-01-26; First posted 2023-02-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Hamstring Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post isometric relaxation (Active Comparator): This Group was treated with baseline treatment of heating for 15min and rehab protocol post isometric relaxation in which 3-5 repetitions for 7-10 seconds hold in each session for three sessions per week in alternate days for four weeks.
  Interventions: Other: Post isometric relaxation
- Post facilitation stretching (Active Comparator): This Group was treated with baseline treatment of heating for 15min and rehab protocol post facilitation stretching in which 3-5 repetitions for 7-10 seconds hold in each session for three sessions per week in alternate days for four weeks.
  Interventions: Other: Post facilitation stretching

INTERVENTIONS:
Other: Post isometric relaxation — post isometric relaxation in which 3-5 repetitions for 7-10 seconds hold in each session for three sessions per week in alternate days for four weeks.
  Arms: Post isometric relaxation
Other: Post facilitation stretching — post facilitation stretching in which 3-5 repetitions for 7-10 seconds hold in each session for three sessions per week in alternate days for four weeks.
  Arms: Post facilitation stretching

SUMMARY:
The goal of this randomized clinical trial is to check the effectiveness of post isometric relaxation and post facilitation stretching on hamstring muscle flexibility in collegiate athletes.

The main question it aims to answer is:

* To compare the post isometric relaxation and post facilitation stretching techniques on hamstring muscle flexibility in collegiate athletes Participants were divided in two groups,
* Group-A was treated with baseline treatment of heating for 15min and rehab protocol post isometric relaxation in which 3-5 repetitions for 7-10 seconds hold in each session for three sessions per week in alternate days for four weeks.
* Group-B was treated with baseline treatment of heating for 15min and rehab protocol post facilitation in which 3-5 repetitions for 7-10 seconds hold in each session for three sessions per week in alternate days for four weeks.

DETAILED DESCRIPTION:
Hamstring injuries are most common injuries in sports and there are many treatment methods and rehabilitation protocols available which are used according to the extent of injury. The main purpose of this study was to check the effectiveness of two treatment techniques on the hamstring muscle flexibility in collegiate athletes. Muscle Energy Techniques (MET) and their related post-isometric relaxation and post facilitation stretching techniques have demonstrated better results in improving flexibility of the tightened muscles. The study was a randomized clinical trial at Pakistan sports board and coaching center Lahore in which convenience sampling technique was used. This study included total 48 participants and for this purpose Open Epi tool software was used as a sample size calculation. Participants falling in this category were recruited into the study, those were male athletes with ages 18 to 35 having bilateral hamstring muscle tightness and acute hamstring injuries. Participants failing to fall in this category were excluded of the study such as females and athletes with hip, buttock and low back pain radiating to back of thigh and history of fractures within 6 months. Universal goniometer, SLR, active knee extension test and sit to reach test would be used as a tool for pre and post assessment of athletes. In this study the subjects were assigned through convenience sampling into two groups. Group A was treated with post isometric relaxation technique and group B was treated with post facilitation technique. Data will analyze through SPSS version 25.0

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 to 35

  * Male
  * Athletes with hamstring muscle tightness (bilateral) or Acute hamstring injuries

Exclusion Criteria:

* • Athletes with hip, buttocks and low back pain radiating to back of thigh

  * History of fracture within 6 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Straight leg raise test. ("change" is being assessed) | Change from Baseline range of motion at 4 weeks
  Straight leg raise (SLR) is a fundamental maneuver during the physical examination of a patient with lower back pain. The straight leg raise test is performed with the patient in a supine position. The examiner gently raises the patient's leg by flexing the hip with the knee in extension, and the test is considered positive when the patient experiences pain along the lower limb in the same distribution of the lower radicular nerve roots (usually L5 or S1)
The sit to reach test ("change" is being assessed) | Change from Baseline range of motion at 4 weeks
  The sit and reach test is a common measure of flexibility, and specifically measures the flexibility of the lower back and hamstring muscles. The starting position for the SR test places the subject's feet against the box relative to the 38.1cm point. After the reach position of the test, the criterion score is 38.1cm plus or minus the distance reached during the test.
The Active Knee Extension Test ("change" is being assessed) | Change from Baseline range of motion at 4 weeks
  The Active Knee Extension Test is used to assess hamstring muscle length and the range of active knee extension in the position of hip flexion. The AKE test subjects were positioned so that the thigh was in contact with the crossbar on the wooden frame apparatus, and the thigh was a t a 90" angle (as measured with the universal goniometer) with the trunk. Subjects were told to extend their knee while maintaining contact with the crossbar.

SECONDARY OUTCOMES:
The Lower Extremity Functional Scale | 4 weeks of intervention
  The Lower Extremity Functional Scale is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. It is efficient to administer and score and is applicable for research purposes and clinical decision making for individual patients. Its maximum score is 80. The lower the score the greater the disability.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiz Zohaib Ahmed, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan sports board Lahore, Lahore, Punjab Province, Pakistan